CLINICAL TRIAL: NCT01384877
Title: A Randomized Double Blind Placebo Controlled Crossover Trial of the Use of Subcutaneous Lidocaine Infusion (SCLI) for Chronic Cancer-related Pain
Brief Title: Subcutaneous Lidocaine For Cancer-Related Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: BC Cancer Foundation (Other)
Responsible Party: Principal Investigator, Pippa Hawley, Palliative Medicine Specialist, British Columbia Cancer Agency
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: H10-00150
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-04

CONDITIONS: Cancer-related Pain
Keywords: Pain; Cancer; Lidocaine; Sodium Channel Blockers
MeSH Terms: conditions — Cancer Pain; Pain; Neoplasms | interventions — Lidocaine; Glucose; Water

STUDY DESIGN:
Intervention Model Description: One-sided McNemar's tests will be carried out to test whether a single infusion of subcutaneous lidocaine will cause a reduction in cancer pain for both the interim and final analyses at the p-values of 0.00153 and 0.02347 respectively.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind performed by pharmacy. Un blinding to occur at end of study. All subjects to be injected with 1 mL of 1% lidocaine subcutaneous prior to the initiation of the study med infusion, which will act as a masking agent.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Experimental): Lidocaine
  Interventions: Drug: Lidocaine
- Placebo (D5W) (Placebo Comparator): Placebo first as compared with lidocaine first
  Interventions: Drug: Placebo (D5W)

INTERVENTIONS:
Drug: Lidocaine — 10mg/kg by subcutaneous infusion over 5.5 hours
  Other Names: Xylocaine; Lignocaine
  Arms: Lidocaine
Drug: Placebo (D5W) — Same volume as for lidocaine infusion, identical clear liquid in appearance, given in same device over same time period (5.5 hrs)
  Other Names: 5% dextrose in water
  Arms: Placebo (D5W)

SUMMARY:
This study's primary objective is to test the hypothesis that a single infusion of subcutaneous lidocaine can cause a clinically useful reduction in cancer pain within 48 hours of infusion and lasting a minimum of 7 days. A clinically useful reduction in pain is defined by either a 2-point reduction (on a 0-10 scale) in the worst pain experienced over a 24-hour period, or a ≥30% reduction in 24-hour opioid requirement. We will use a composite endpoint of reduction in pain without increase in 24-hr opioid requirement or no decrease in pain with a ≥30% reduction in 24-hour opioid requirement.Subjects will receive either lidocaine or placebo, followed at least 1 week later by the alternate agent.

DETAILED DESCRIPTION:
Ten mg/kg of lidocaine will be infused subcutaneously via a Baxter infusor over a 5.5 hour period in ambulatory adult cancer patients with a worst pain score of at least 4 out of 10 despite therapy with at least one opioid plus appropriate oral adjuvant analgesic(s).

A clinically useful reduction in pain is defined by either a 2-point reduction (on a 0-10 scale) in the worst pain experienced over a 24-hour period, or a ≥30% reduction in 24-hour opioid requirement.

The secondary objectives are 1) to determine whether any significant toxicities occur as a result of the infusion. For this study significant toxicity is considered as any adverse event which either leads to the infusion being terminated, or which leads to medical intervention, such as prescribing of another medication or equivalent treatment, 2) to determine the effect of Lidocaine infusion on QOL parameters as measured by the Patient Outcome Scale (POS) Questionnaire and 3) to determine the duration of response to lidocaine infusion.

Subjects will fill out Brief Pain Inventory (BPI), Patient Outcome Scale (POS) periodically and medication logs daily while on study.

On Days of treatment the subjects will have vital sign monitoring every 15 minutes for the 1st hour and then periodically as set out in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years of age or older
* In or outpatients referred to the BCCA PSMPC Clinics with a diagnosis of cancer
* Subjects must have somatic, visceral or neuropathic pain related to cancer
* Pain intensity, measured by a worst pain score over the last 72 hours of ≥4 on a 0-10 numerical rating scale
* Must have tried at least one opioid medication without adequate response or with significant side-effects for at least one week
* For those with neuropathic pain, must have also tried at least one adjuvant analgesic, such as a tricyclic (unless contraindicated) or an anticonvulsant without adequate response or with significant side-effects for at least one week
* Life expectancy of > 3 months
* Must be able to communicate symptoms indicating potential toxicity of Lidocaine
* Must have a competent caregiver in the home overnight after each infusion
* Must be willing to remain within 30 minutes of the Cancer Centre during each infusion

Exclusion Criteria:

* Clinically significant cardiac disease, i.e, cardiac failure, atrial fibrillation with slow ventricular rate (<60), any degree of heart block
* New analgesic treatment initiated in time frame which might have effect within one week of study drug.
* Hyper or hypokalemia.
* Liver failure (bilirubin ≥ 25 umol/L).
* Renal failure (eGFR <50% of normal)
* Uncontrolled hypertension (>160/90).
* Hypotension (systolic < 90).
* Uncontrolled seizures.
* Planned initiation of chemotherapy, radiotherapy or bisphosphonates within 30 days prior to treatment with study drug.
* Received an investigational drug within 30 days prior to study.
* History of allergy to lidocaine or other topical, local or infusional anesthetics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-12; Primary Completion 2017-12 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippa H Hawley, B.Med, FRCPC, Principal Investigator — British Columbia Cancer Agency
Locations (2):
- Canada (2):
  - BC Cancer Center of the North, Prince George, British Columbia
  - BC Cancer Agency, Vancouver, British Columbia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One (1) participant signed the informed consent form but withdrew from the study before receiving any treatment.
Groups:
- Lidocaine/Placebo: Patient received Lidocaine in the first period followed by placebo in the second period.
  Lidocaine: 10mg/kg by subcutaneous infusion over 5.5 hours
  Placebo (D5W): Same volume as for lidocaine infusion, identical clear liquid in appearance, given in same device over 5.5 hrs
- Placebo (D5W)/Lidocaine: Patient received Placebo in the first period followed by Lidocaine in the second period.
  Placebo (D5W): Same volume as for lidocaine infusion, identical clear liquid in appearance, given in same device over 5.5 hrs
  Lidocaine: 10mg/kg by subcutaneous infusion over 5.5 hours
Period: Treatment 1
Arm/Group | Lidocaine/Placebo | Placebo (D5W)/Lidocaine
Started | 17 | 15
Completed | 17 | 15
Not Completed | 0 | 0
Period: Treatment 2
Arm/Group | Lidocaine/Placebo | Placebo (D5W)/Lidocaine
Started | 16 (1 Patient died between treatment periods) | 13 (2 Patients died between treatment periods)
Completed | 14 | 11
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: The overall number in the baseline analysis include all participants who signed the informed consent form. One (1) participant included in this analysis withdrew before receiving any treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine/Placebo | Placebo (D5W)/Lidocaine | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 10 | 7 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 17 | 16 | 33
Palliative Performance Scale [Count of Participants; unit: Participants] — Palliative Performance Scale (PPS) PPS ranges from 100% to 0%
  100%: Patient has full ambulation; normal activity and work; no evidence of disease; full self-care; normal intake; full conscious level
  50%: Patient mainly sit/lie; unable to do any work; extensive disease; considerable assistance required for self-care; normal or reduced intake; full or confusion level of consciousness
  0% death
  Participants
    100% | 1 | 0 | 1
    90-99% | 6 | 4 | 10
    80-89% | 1 | 0 | 1
    70-79% | 8 | 8 | 16
    60-69% | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reduction in Worst Pain Intensity or Reduction in 24hr Opioid Dose of at Least 30% Without Worsening of Pain Scores
Description: The primary outcomes measure is a binary variable indicating whether lidocaine caused a reduction in cancer pain within 48 hours of infusion and lasting a minimum of 7 days. Lidocaine will be considered to have caused reduction in cancer pain if the subject had either one of the following episodes and lasting a minimum of 7 days:
  1. A 2-point reduction in severity of pain as assessed by the worst pain score in the last 24 hours (question 3) of the Brief Pain Inventory - Short Form (BPI), compared to the BPI pain score at baseline.
     Or:
  2. ≥30% reduction in 24-hour opioid dose.
Time Frame: 7 days
Population: Participants were included in analysis if they completed both treatment periods and all the data was collected for both treatment periods
Measure: Count of Participants; unit: Participants
Arm/Group | Lidocaine/Placebo | Placebo (D5W)/Lidocaine
Number analyzed (Participants) | 14 | 11
Participants
  Period 1 | 1 | 2
  Period 2 | 2 | 1

2. Secondary Outcome: Quality of Life Question: Over the Past 3 Days, Have You Been Affected by Pain?
Description: Effect of Lidocaine infusion on Quality Of Life parameters as measured by the Patient Outcome Scale (POS) Questionnaire Baseline scores were compared to an average post treatment score (taken immediately post treatment and on days 2, 3, and 7 following treatment) All POS questions were scored from 0 to 4 with lower scores requiring less clinical attention than higher scores
Time Frame: At most 6 weeks (duration of study)
Population: Participants included in this analysis completed both treatment periods and returned all their questionnaires at the end of the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine/Placebo | Placebo (D5W)/Lidocaine
Number analyzed (Participants) | 15 | 12
score on a scale
  Baseline | 2.93 (0.59) | 2.67 (0.65)
  Period 1 | 2.62 (.041) | 2.52 (0.47)
  Period 2 | 2.52 (0.54) | 2.40 (0.60)

3. Secondary Outcome: Quality of Life Question: Over the Past 3 Days, Have Other Symptoms e.g. Feeling Sick, Having a Cough or Constipation Been Affecting How You Feel?
Description: as for outcome 2
Time Frame: At most 6 weeks (duration of study)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine/Placebo | Placebo (D5W)/Lidocaine
Number analyzed (Participants) | 15 | 12
score on a scale
  Baseline | 1.47 (1.36) | 1.5 (0.8)
  Period 1 | 1.40 (0.68) | 1.29 (0.79)
  Period 2 | 1.43 (1.79) | 0.95 (0.82)

4. Secondary Outcome: Quality of Life Question: Over the Past 3 Days, Have You Been Feeling Anxious or Worried About Your Illness or Treatment?
Description: as for outcome 2
Time Frame: At most 6 weeks (duration of study)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine/Placebo | Placebo (D5W)/Lidocaine
Number analyzed (Participants) | 15 | 12
score on a scale
  Baseline | 2.13 (0.92) | 1.67 (1.07)
  Period 1 | 1.92 (0.67) | 1.71 (0.8)
  Period 2 | 1.73 (0.68) | 1.47 (0.83)

5. Secondary Outcome: Quality of Life Question: Over the Past 3 Days, Have Any of Your Family or Friends Been Anxious or Worried About You?
Description: as for outcome 2
Time Frame: At most 6 weeks (duration of study)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine/Placebo | Placebo (D5W)/Lidocaine
Number analyzed (Participants) | 15 | 12
score on a scale
  Baseline | 1.60 (0.91) | 1.67 (1.07)
  Period 1 | 1.53 (0.72) | 1.71 (1.06)
  Period 2 | 1.50 (0.62) | 1.45 (1.12)

6. Secondary Outcome: Quality of Life Question: Over the Past 3 Days, Have You Been Able to Share How You Are Feeling With Your Family or Friends?
Description: as for outcome 2
Time Frame: At most 6 weeks (duration of study)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine/Placebo | Placebo (D5W)/Lidocaine
Number analyzed (Participants) | 15 | 12
score on a scale
  Baseline | 0.87 (1.06) | 1.33 (1.07)
  Period 1 | 1.27 (1.04) | 1.32 (1.10)
  Period 2 | 1.12 (1.06) | 1.50 (1.44)

7. Secondary Outcome: Quality of Life Question: Over the Past 3 Days, Have You Been Feeling Depressed?
Description: as for outcome 2
Time Frame: At most 6 weeks (duration of study)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine/Placebo | Placebo (D5W)/Lidocaine
Number analyzed (Participants) | 15 | 12
score on a scale
  Baseline | 1.67 (1.05) | 1.25 (1.14)
  Period 1 | 1.55 (1.00) | 1.55 (0.97)
  Period 2 | 1.46 (0.83) | 1.23 (0.96)

8. Secondary Outcome: Quality of Life Question: Over the Past 3 Days, Have You Felt Good About Yourself as a Person?
Description: as for outcome 2
Time Frame: At most 6 weeks (duration of study)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine/Placebo | Placebo (D5W)/Lidocaine
Number analyzed (Participants) | 15 | 12
score on a scale
  Baseline | 1.73 (0.96) | 1.75 (1.22)
  Period 1 | 1.73 (0.94) | 1.52 (1.02)
  Period 2 | 1.78 (1.05) | 1.37 (1.05)

9. Secondary Outcome: Quality of Life Question: Over the Past 3 Days, How Much Time do You Feel Has Been Wasted on Appointments Relating to Your Healthcare e.g. Waiting Around for Transport or Repeating Tests?
Description: as for outcome 2
Time Frame: At most 6 weeks (duration of study)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine/Placebo | Placebo (D5W)/Lidocaine
Number analyzed (Participants) | 15 | 12
score on a scale
  Baseline | 0.67 (1.23) | 0.50 (1.24)
  Period 1 | 0.65 (1.00) | 0.77 (0.97)
  Period 2 | 0.55 (0.87) | 0.43 (0.60)

10. Secondary Outcome: Quality of Life Question: Over the Past 3 Days, Have Any Practical Matters Resulting From Your Illness, Either Financial or Personal, Been Addressed?
Description: as for outcome 2
Time Frame: At most 6 weeks (duration of study)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lidocaine/Placebo | Placebo (D5W)/Lidocaine
Number analyzed (Participants) | 15 | 12
score on a scale
  Baseline | 1.08 (1.04) | 1.0 (1.35)
  Period 1 | 1.17 (1.44) | 1.12 (1.29)
  Period 2 | 1.20 (1.41) | 0.93 (1.29)

ADVERSE EVENTS:
Time Frame: 21 days after each treatment, up to 6 weeks total
Arm/Group | Lidocaine | Placebo (D5W)
All-Cause Mortality (participants affected / at risk) | 1/32 | 2/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 3/32 | 2/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine (N=32) | Placebo (D5W) (N=32)
Tingling (Nervous system disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Feet Swollen (General disorders) | 1 (2) | 0 (0)
Throbbing sensation from waist down (Nervous system disorders) | 1 (1) | 0 (0)
Neck Hurts (General disorders) | 1 (2) | 0 (0)
Blood in Urine (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) — above right hip going up back and down leg
Fatigue (General disorders) | 1 (2) | 0 (0)
Swelling at needle site (General disorders) | 1 (1) | 0 (0)
Redness at needle site (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT01384877/Prot_SAP_000.pdf